CLINICAL TRIAL: NCT02185664
Title: Comparison of the Landmark Technique and the Static Ultrasound Guided Technique for Internal Jugular Vein Cannulation in Adult Cardiac Surgical Patients.
Brief Title: Use of Static Ultrasound Guidance for Internal Jugular Vein Cannulation in Adult Cardiac Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Deepti Saigal, Assistant Professor, Govind Ballabh Pant Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: F.2/IEC/MAMC/11/No.96
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Adult Cardiac Surgical Patients
Keywords: internal jugular vein; landmark; ultrasound; static; cardiac surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Landmark technique (Active Comparator): The landmark technique is the standard technique used for internal jugular vein cannulation.
  Interventions: Procedure: landmark technique
- Static Ultrasound technique (Experimental): Static ultrasound technique was used to assist internal jugular vein cannulation.
  Interventions: Device: Static Ultrasound technique

INTERVENTIONS:
Procedure: landmark technique — The apex of the imaginary triangle formed between the two heads of sternocleidomastoid and clavicle was used as the point of needle entry, just lateral to the pulsation of the internal carotid artery and directed towards the ipsilateral nipple at an angle of 45 degrees.
  Arms: Landmark technique
Device: Static Ultrasound technique — Static ultrasound guided internal jugular vein cannulation was performed by using the transthoracic echocardiography probe supplied with the transesophageal echocardiography machine in the cardiothoracic surgery operation theatre. The internal jugular vein was located and marked using this method prior to puncture.
  Arms: Static Ultrasound technique

SUMMARY:
Cannulation of the internal jugular vein (IJV) for central venous access is a standard practice in cardiac surgery. In this study, the authors tested the hypothesis that using an ultrasound (US) scanner would increase the success of IJV cannulation and decrease the incidence of complications in adult cardiac surgical patients.

The study will include adult cardiac surgical patients, randomized into two groups (control vs. US). In the control group, IJV cannulation will be performed by the conventional landmark technique using Seldinger method. In the US group, the course of the IJV will be marked before cannulation using a 2 - 4 MHz transthoracic echocardiography probe. The success rate, number of attempts, cannulation time and complication rate will be compared for the two groups.

DETAILED DESCRIPTION:
Use of real time ultrasound has recently been recommended as the standard of care for insertion of central venous catheters. However, its usage is limited by various factors which include availability, space constraints and perceived lack of need according to surveys including cardiovascular anesthesiologists. We will conduct a prospective randomized controlled trial to compare the conventional landmark technique with the static ultrasound (US) technique that utilized the transthoracic echocardiography (TTE) ultrasound probe which is supplied along with the transesophageal echocardiography machines for internal jugular vein cannulation in adult cardiac surgical patients.

After ethical committee approval and patient consent, adult patients scheduled for elective cardiac surgery will be randomized to undergo internal jugular vein cannulation by either of the two methods: standard landmark technique (group A: control group), static US technique using the TTE probe (group B: ultrasound group). The success rate, number of attempts, total cannulation time and complication rate in the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for elective cardiac surgery

Exclusion Criteria:

* patients undergoing bidirectional Glenn shunt, Fontan surgery or emergency surgery
* local site infection
* presence of coagulopathy
* anatomical deformity of neck(burns, neck swelling, surgical scar)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
success | during internal jugular venous cannulation
  Success was defined as location of the IJV by the finder needle within five attempts.

SECONDARY OUTCOMES:
number of attempts by finder/locator needle | at the time of internal jugular vein cannulation
  The total number of attempts taken to locate the internal jugular vein using the locator/finder needle were measured.
total number of attempts by puncture needle | at the time of internal jugular vein cannulation
  The total number of attempts taken by the puncture needle to enter the internal jugular vein were measured.
First attempt sucess | at the time of internal jugular vein cannulation
  First attempt success was defined as location of the IJV by finder needle in the first attempt.
Central venous cannulation time | at the time of internal jugular venous cannulation
  Time to central venous cannulation (CVC) was defined as the time taken from the insertion of finder needle till de-airing and flushing of all the three ports of the triple lumen catheter.
ultrasound time | at the time of internal jugular vein cannulation
  The duration of ultrasound was defined as the time between the placement of the probe on neck till the marking of the course of the vein on the skin.
total cannulation time | at the time of internal jugular vein cannulation
  control group: total cannulation time= central venous cannulation time ultrasound group: total cannulation time= central venous cannulation time+ ultrasound time
complication rate | at the time of central venous cannulation
  The complication rate was calculated as a percentage of the total number of complications with respect to the sample size

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Tempe, MD, Principal Investigator — Govind Ballabh pant Hospital and Maulana azad Medical College, New Delhi, India
Locations (1):
- Department of Anesthesia and Intensive Care, Govind Ballabh Pant Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Espinet A, Dunning J. Does ultrasound-guided central line insertion reduce complications and time to placement in elective patients undergoing cardiac surgery. Interact Cardiovasc Thorac Surg. 2004 Sep;3(3):523-7. doi: 10.1016/j.icvts.2004.05.006. PMID 17670301
- [Background] Bailey PL, Glance LG, Eaton MP, Parshall B, McIntosh S. A survey of the use of ultrasound during central venous catheterization. Anesth Analg. 2007 Mar;104(3):491-7. doi: 10.1213/01.ane.0000255289.78333.c2. PMID 17312193
- [Result] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984